CLINICAL TRIAL: NCT00947349
Title: Safety, Pharmacokinetics and Antiviral Effect of BI 201335 NA in HCV-1 Infected Patients Treated for 28 Days for Treatment naïve and Experienced Patients Treated in Combination With Peg Interferon Alfa-2a and Ribavirin
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 201335 as Softgel Capsule in Naive Hepatitis C Virus (HCV) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.14
Record Dates: First submitted 2009-07-21; First posted 2009-07-28 (Estimated); Results first posted 2015-07-07 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C; Pharmacokinetics
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

ARMS (4):
- BI 201335 NA low TN (Experimental): patient to receive a capsule containing low dose of BI 201335 NA/Drug for treatment-naive (TN) patients
  Interventions: Drug: pegylated interferon (PegIFN) alfa-2a; Drug: BI 201335 NA low placebo; Drug: ribavirin (RBV); Drug: BI 201335 NA low
- BI 201335 NA high TN (Experimental): patient to receive a capsule containing high dose of BI 201335 NA/Drug for treatment-naive (TN )patients
  Interventions: Drug: ribavirin (RBV); Drug: pegylated interferon (PegIFN) alfa-2a; Drug: BI 201335 NA high; Drug: BI 201335 NA high placebo
- BI 201335 NA high TE (Experimental): patient to receive a capsule containing high dose of BI 201335 NA/Drug for treatment-experienced (TE) patients
  Interventions: Drug: pegylated interferon (PegIFN) alfa-2a; Drug: ribavirin (RBV); Drug: BI 201335 NA high
- Placebo in Treatment Naive (TN) Patients (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ribavirin (RBV) — ribavirin (RBV)
  Arms: BI 201335 NA high TN
Drug: pegylated interferon (PegIFN) alfa-2a — pegylated interferon (PegIFN) alfa-2a
  Arms: BI 201335 NA low TN
Drug: pegylated interferon (PegIFN) alfa-2a — pegylated interferon (PegIFN) alfa-2a
  Arms: BI 201335 NA high TE
Drug: ribavirin (RBV) — ribavirin (RBV)
  Arms: BI 201335 NA high TE
Drug: BI 201335 NA low placebo — Placebo
  Arms: BI 201335 NA low TN
Drug: pegylated interferon (PegIFN) alfa-2a — pegylated interferon (PegIFN) alfa-2a
  Arms: BI 201335 NA high TN
Drug: ribavirin (RBV) — ribavirin (RBV)
  Arms: BI 201335 NA low TN
Drug: BI 201335 NA high — BI 201335 NA high
  Arms: BI 201335 NA high TN
Drug: BI 201335 NA low — BI 201335 NA
  Arms: BI 201335 NA low TN
Drug: BI 201335 NA high placebo — placebo
  Arms: BI 201335 NA high TN
Drug: BI 201335 NA high — BI 201335 NA high
  Arms: BI 201335 NA high TE
Drug: Placebo
  Arms: Placebo in Treatment Naive (TN) Patients

SUMMARY:
The current Standard of Care (SOC) for chronic HCV infection, which is pegylated interferon-alfa as combination therapy with ribavirin for 24-48 weeks of treatment, is effective in only part of the patients and is often associated with severe adverse effects leading to discontinuation of treatment and dose modifications.

A number of compounds with direct activity are currently under clinical development, incl. BI 201335. BI 201335 works by preventing the Hepatitis C virus from replicating by binding to the HCV protease (enzyme). The main purpose of this clinical trial with BI 201335 is to see how well BI 201335 works and how safe BI 201335 is to use daily in combination with PegIFN and RBV in HCV infected patients

ELIGIBILITY:
Inclusion criteria:

* chronic HCV genotype-1;
* high viral load

Exclusion criteria:

* Mixed genotype (1/2, 1/3, or 1/4), diagnosed by genotypic testing at screening
* Previous treatment with protease inhibitor

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Japan (3):
  - 1220.14.003 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 1220.14.001 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 1220.14.002 Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo in Treatment Naive (TN) Patients: Matching placebo to BI 201335 (Faldaprevir) NA (sodium) with PegIFN/RBV in TN patients
- BI 201335 NA Low for Treatment Naive (TN): Patients receive a capsule containing low dose of BI 201335 NA (120 mg q.d. (once daily)) with PegIFN/RBV in treatment naive (TN) patients
- BI 201335 NA High TN: Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV in TN patients
- BI 201335 NA High for Treatment Experienced (TE): Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV in treatment experienced (TE) patients.
Period: Triple Treatment Combination Period
Arm/Group | Placebo in Treatment Naive (TN) Patients | BI 201335 NA Low for Treatment Naive (TN) | BI 201335 NA High TN | BI 201335 NA High for Treatment Experienced (TE)
Started | 4 | 6 | 6 | 6
Completed | 4 | 5 | 6 | 6
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Overall Study Standard of Care
Arm/Group | Placebo in Treatment Naive (TN) Patients | BI 201335 NA Low for Treatment Naive (TN) | BI 201335 NA High TN | BI 201335 NA High for Treatment Experienced (TE)
Started | 4 | 5 | 6 | 6
Completed | 4 | 5 | 4 | 4
Not Completed | 0 | 0 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consisted of all patients who were given study medication and were documented to have taken at least one dose of investigational products regardless of randomisation.
Groups:
- Placebo in TN Patients: Matching placebo to BI 201335 NA with PegIFN/RBV in TN patients
- BI 201335 NA Low TN: Patients receive a capsule containing low dose of BI 201335 NA (120 mg q.d.) with PegIFN/RBV in TN patients
- BI 201335 NA High TN: Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.). with PegIFN/RBV in TN patients
- BI 201335 NA High TE: Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV in TE patients
- Total: Total of all reporting groups
Arm/Group | Placebo in TN Patients | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE | Total
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (6.0) | 48.0 (13.5) | 56.0 (9.2) | 58.0 (8.3) | 53.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 0 | 9
  Male | 3 | 2 | 2 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Investigator Defined Drug-related Adverse Events in Triple Combination Therapy
Description: Drug-related AEs were defined as those whose causal relationship with any one of the investigational products was considered by the investigator.
Time Frame: 4 weeks
Population: The treated set (TS) consisted of all patients who were given study medication and were documented to have taken at least one dose of investigational products regardless of randomization randomisation.
Measure: Number; unit: participants
Groups:
- Triple TN Placebo: Triple combination therapy for treatment naive patients- Patients receive a capsule containing matching placebo to BI 201335 NA (Placebo with PegIFN/RBV).
- Triple TN 120 mg: Triple combination therapy for treatment naive patients- Patients receive a capsule containing low dose of BI 201335 NA (120 mg q.d.) with PegIFN/RBV.
- Triple TN 240 mg: Triple combination therapy for treatment naive patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV.
- Triple TE 240 mg: Triple combination therapy for treatment experienced patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV.
Arm/Group | Triple TN Placebo | Triple TN 120 mg | Triple TN 240 mg | Triple TE 240 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 3 | 6 | 6 | 5

2. Primary Outcome: Number of Patients With Possible Clinically Significant Laboratory Abnormalities in Triple Combination Therapy
Description: Frequency of patients with possible clinically significant abnormalities or clinically significant laboratory test value changes over time in triple combination therapy for treatment naive patients and treatment experienced patients.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Triple TN Placebo | Triple TN 120 mg | Triple TN 240 mg | Triple TE 240 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants
  Decrease Haematocrit | 2 | 2 | 3 | 4
  Decrease Haemoglobin | 3 | 3 | 2 | 4
  Decrease Red blood cell ct. | 1 | 2 | 2 | 2
  Decrease White blood cell ct. | 2 | 4 | 5 | 4
  Decrease Platelets | 0 | 1 | 0 | 0
  Increase Eosinophils | 0 | 0 | 1 | 0
  Decrease Sodium | 1 | 2 | 2 | 1
  Decrease Potassium | 0 | 0 | 1 | 0
  Decrease Bicarbonate | 0 | 1 | 0 | 1
  Increase Bicarbonate | 1 | 2 | 1 | 2
  Increase Bilirubin, total | 0 | 2 | 6 | 5
  Increase Bilirubin, direct | 0 | 1 | 3 | 4
  Increase Protein, total | 0 | 0 | 1 | 0
  Increase Uric acid | 2 | 2 | 0 | 1
  Increase Triglyceride | 0 | 0 | 1 | 4
  Increase U. pH | 0 | 1 | 0 | 0

3. Secondary Outcome: Week 2 Virological Response (W2VR)
Description: Number of patients satisfying W2VR (plasma HCV RNA (Hepatitis C Virus Ribonucleic acid) level below the limit of quantification (BLQ))
Time Frame: 2 weeks
Population: The full analysis set (FAS) consisted of all randomised patients who were given investigational products and were documented to have taken at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- Placebo in TN: Matching placebo to BI 201335 NA with PegIFN/RBV in TN patients
Arm/Group | Placebo in TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 0 | 5 | 6 | 3

4. Secondary Outcome: Week 4 Virological Response (W4VR)
Description: Number of patients satisfying W4VR (plasma HCV RNA level below the limit of quantification (BLQ))
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Groups:
- Placebo TN: Matching placebo to BI 201335 NA with PegIFN/RBV in TN patients
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 0 | 6 | 6 | 5

5. Secondary Outcome: Rapid Virological Response (RVR)
Description: Number of patients satisfying RVR (plasma HCV RNA level below the limit of detection (BLD) at Week 4)
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 0 | 5 | 6 | 4

6. Secondary Outcome: Change From Baseline in HCV Viral Load
Description: Change form baseline in HCV viral load (log10) after 4 weeks
Time Frame: baseline and week 4
Population: as for outcome 3
Measure: Mean (Standard Error); unit: IU/mL
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
IU/mL | -3.30 (0.74) | -5.88 (0.17) | -5.95 (0.21) | -5.53 (0.29)

7. Secondary Outcome: Day 28 Virologic Response
Description: Number of patients with HCV viral load reduction >= 2 log10 at Week 4
Time Frame: 4 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 3 | 6 | 6 | 6

8. Secondary Outcome: Early Virological Response (EVR)
Description: Number of patients with reduction >= 2 log10 in plasma HCV RNA level at Week 12
Time Frame: 12 Weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 4 | 5 | 6 | 6

9. Secondary Outcome: Complete Early Virological Response (cEVR)
Description: Number of patients with plasma HCV RNA level BLD at Week 12
Time Frame: 12 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 3 | 5 | 5 | 6

10. Secondary Outcome: End of Treatment Response (ETR)
Description: Number of patients with plasma HCV RNA level BLD at week 48
Time Frame: 48 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 3 | 5 | 4 | 4

11. Secondary Outcome: Sustained Virologic Response (SVR)
Description: Number of patients with plasma HCV RNA level BLD 24 weeks after treatment completion
Time Frame: 72 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants | 2 | 4 | 5 | 3

12. Secondary Outcome: Number of Participants With Investigator Defined Drug-related Adverse Events in Standard of Care (SOC) With PegIFN α-2a and RBV
Description: Drug-related AEs in SOC treatment period were defined as those whose causal relationship with any one of the investigational products was considered by the investigator.
Time Frame: 44 weeks
Population: as for baseline characteristics
Measure: Number; unit: participant(s)
Groups:
- SOC TN Placebo: Standard of care (SOC) for treatment naive patients- Patients receive a capsule containing matching placebo to BI 201335 NA (Placebo with PegIFN/RBV).
- SOC TN 120 mg: Standard of care for treatment naive patients- Patients receive a capsule containing low dose of BI 201335 NA (120 mg q.d.) with PegIFN/RBV.
- SOC TN 240 mg: Standard of care for treatment naive patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV.
- SOC TE 240 mg: Standard of care for treatment experienced patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with PegIFN/RBV.
Arm/Group | SOC TN Placebo | SOC TN 120 mg | SOC TN 240 mg | SOC TE 240 mg
Number analyzed (Participants) | 4 | 5 | 6 | 6
participant(s) | 3 | 5 | 4 | 5

13. Secondary Outcome: Number of Patients With Possible Clinically Significant Laboratory Abnormalities in Standard of Care (SOC) With PegIFN α-2a and RBV
Description: Frequency of patients with possible clinically significant abnormalities or clinically significant laboratory test value changes over time in SOC period for treatment naive patients and treatment experienced patients.
Time Frame: 44 weeks
Population: TS
Measure: Number; unit: participant(s)
Arm/Group | SOC TN Placebo | SOC TN 120 mg | SOC TN 240 mg | SOC TE 240 mg
Number analyzed (Participants) | 4 | 5 | 6 | 6
participant(s)
  Decrease haematocrit | 1 | 3 | 5 | 4
  Decrease haemoglobin | 4 | 2 | 2 | 5
  Decrease red blood cell ct. | 0 | 3 | 4 | 3
  Decrease white blood cell ct. | 3 | 5 | 5 | 3
  Decrease platelets | 0 | 1 | 0 | 0
  Increase eosinophils | 0 | 0 | 1 | 1
  Decrease sodium | 1 | 0 | 1 | 0
  Decrease potassium | 0 | 0 | 1 | 0
  Increase bicarbonate | 0 | 1 | 0 | 0
  Increase uric acid | 1 | 0 | 0 | 0
  Increase triglyceride | 1 | 0 | 0 | 2
  Increase U. pH | 0 | 2 | 0 | 0
  Increase AST/GOT, SGOT | 0 | 1 | 0 | 1
  Increase ALT/GPT, SGPT | 0 | 1 | 0 | 1

14. Secondary Outcome: Assessment of Tolerability in Standard of Care (SOC) With PegIFN α -2a and RBV
Description: An assessment of tolerability for the safety of the SOC with PegIFN alfa-2a and RBV.
Time Frame: 44 weeks
Population: TS
Measure: Number; unit: participant(s)
Arm/Group | SOC TN Placebo | SOC TN 120 mg | SOC TN 240 mg | SOC TE 240 mg
Number analyzed (Participants) | 4 | 5 | 6 | 6
participant(s)
  Good | 2 | 4 | 1 | 3
  Satisfactory | 2 | 0 | 2 | 1
  Not satisfactory | 0 | 1 | 1 | 2
  Bad | 0 | 0 | 2 | 0

15. Secondary Outcome: AUCτ,1 for BI 201335 ZW
Description: Area under the curve (AUC) concentration after the first dose of BI 201335 ZW
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the first dose
Population: The pharmacokinetic analysis set (PKS) consisted of all randomised patients who took at least one dose of investigational products and with at least one on treatment blood sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 6 | 4 | 6
ng*h/mL | 68900 (25.3) | 171000 (21.2) | 233000 (38.5)

16. Secondary Outcome: Cmax of BI 201335 ZW
Description: Maximum concentration of BI 201335 ZW after multiple oral admin. of BI 201335 NA with RBV and PegIFN alfa-2a
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the first dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 6 | 4 | 6
ng/mL | 5500 (24.4) | 12600 (29.0) | 15000 (40.0)

17. Secondary Outcome: AUCτ,ss of BI 201335 ZW
Description: AUC at steady state after 4 weeks combination of the last dose
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
ng*h/mL | 70800 (86.5) | 361000 (68.0) | 499000 (41.3)

18. Secondary Outcome: Cmax,ss of BI 201335 ZW
Description: Maximum concentration of BI 201335 ZW at steady state
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
ng/mL | 5880 (61.5) | 24500 (52.2) | 29100 (35.3)

19. Secondary Outcome: AUCτ,1 for Ribavirin (RBV)
Description: Area under the plasma concentration curve of RBV after the first dose of placebo or BI 201335 NA with with RBV and PegIFN alfa-2a
Time Frame: -0:10, 1,2,3,4,5,6,8,10,11:50, 23:50 hours on the first dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Placebo TN: Matching placebo to BI 201335 NA with RBV and PegIFN alfa-2a in TN patients
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 4 | 6
ng*h/mL | 5160 (22.1) | 4660 (35.8) | 4620 (22.9) | 3500 (41.2)

20. Primary Outcome: Assessment of Tolerability in Triple Combination Therapy
Description: An assessment of tolerability for the safety of the triple combination therapy with BI 201335 NA, PegIFN α -2a and RBV.
Time Frame: 4 weeks
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Triple TN Placebo | Triple TN 120 mg | Triple TN 240 mg | Triple TE 240 mg
Number analyzed (Participants) | 4 | 6 | 6 | 6
participants
  Good | 3 | 5 | 5 | 6
  Satisfactory | 0 | 1 | 1 | 0
  Not Satisfactory | 1 | 0 | 0 | 0
  Bad | 0 | 0 | 0 | 0

21. Secondary Outcome: Cmax of RBV
Description: Maximum Plasma concentration of RBV after multiple oral admin. of placebo with RBV and PegIFN alfa-2a
Time Frame: -0:10, 1,2,3,4,5,6,8,10,11:50, 23:50 hours on the first dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Placebo TN: Matching placebo to BI 201335 NA with RBV and PegIFN alfa- 2a in TN patients
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 4 | 6
ng/mL | 1130 (24.9) | 761 (29.7) | 724 (33.7) | 509 (51.0)

22. Secondary Outcome: AUCτ,ss of RBV
Description: Area under the plasma concentration curve of RBV after the multiple oral administration of BI 201335 NA (or placebo) with RBV and PegIFN alfa-2a at steady state
Time Frame: -0:10, 1,2,3,4,5,6,8,10,11:50, 23:50 hours on the last dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 5 | 6
ng*h/mL | 27500 (29.5) | 25200 (42.4) | 22400 (38.5) | 20000 (18.7)

23. Secondary Outcome: Cmax,ss of RBV
Description: Maximum Plasma concentration of RBV after multiple oral admin. of BI 201335 NA (or placebo) with RBV and PegIFN alfa-2a at steady state
Time Frame: -0:10, 1,2,3,4,5,6,8,10,11:50, 23:50 hours on the last dose
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 5 | 5 | 6
ng/mL | 3060 (35.4) | 2710 (47.3) | 2280 (43.2) | 2130 (18.0)

24. Secondary Outcome: Tmax for BI 201335 ZW
Description: Time to maximum plasma concentration (tmax) of BI 201335 ZW after the first dose of BI 201335 NA with RBV and PegIFN alfa-2a
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the first dose
Population: PKS
Measure: Median (Full Range); unit: hour(s)
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 6 | 4 | 6
hour(s) | 4.98 [3.92 to 9.88] | 5.50 [4.03 to 7.93] | 7.97 [2.88 to 9.92]

25. Secondary Outcome: Tmax for RBV
Description: Time to maximum plasma concentration (tmax) of RBV after the first dose of BI 201335 NA with RBV and PegIFN alfa-2a
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the first dose
Population: PKS
Measure: Median (Full Range); unit: hour(s)
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 6 | 4 | 6
hour(s) | 1.94 [0.917 to 3.00] | 3.98 [2.00 to 4.88] | 3.92 [2.05 to 5.97] | 4.98 [1.97 to 6.02]

26. Secondary Outcome: Tmax, ss for BI 201335 ZW
Description: Time from last dosing to the maximum plasma concentration (tmax) of BI 201335 ZW after the last dose of BI 201335 NA with RBV and PegIFN alfa-2a at steady state
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Median (Full Range); unit: hour(s)
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
hour(s) | 3.83 [1.85 to 5.07] | 2.99 [2.90 to 3.05] | 3.49 [2.92 to 4.03]

27. Secondary Outcome: Tmax, ss for RBV
Description: Time to the maximum plasma concentration (tmax) of RBV after the last dose of BI 201335 NA with RBV and PegIFN alfa-2a at steady state
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Median (Full Range); unit: hour(s)
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 5 | 5 | 6
hour(s) | 2.42 [0.90 to 3.93] | 2.92 [1.85 to 4.08] | 2.90 [1.93 to 5.88] | 3.92 [2.00 to 5.03]

28. Secondary Outcome: t1/2,ss for BI 201335 ZW
Description: terminal half-life of the analyte in plasma at steady state (t1/2,ss)
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour(s)
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
hour(s) | 29.3 (7.70) | 21.2 (9.00) | 23.0 (19.8)

29. Secondary Outcome: Cmin,ss for BI 201335 ZW
Description: Minimum concentration of the analyte (BI 201335 ZW) in plasma over the dosing interval at steady state
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
ng/mL | 1550 (138) | 10200 (85.0) | 16000 (54.1)

30. Secondary Outcome: Cmin,ss for RBV
Description: Minimum concentration of the analyte (RBV) in plasma over the dosing interval at steady state
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 5 | 5 | 6
ng/mL | 1980 (24.6) | 1730 (44.0) | 1590 (36.4) | 1400 (18.5)

31. Secondary Outcome: Cavg for BI 201335 ZW
Description: average plasma concentration (Cavg) of BI 201335 ZW
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
ng/mL | 2950 (86.5) | 15000 (68.0) | 20800 (41.3)

32. Secondary Outcome: Cavg for RBV
Description: average plasma concentration (Cavg) of RBV
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Placebo TN | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 4 | 5 | 5 | 6
ng/mL | 2290 (29.5) | 2100 (42.4) | 1860 (38.5) | 1670 (18.7)

33. Secondary Outcome: CL/F,ss for BI 201335 ZW
Description: apparent clearance of the analyte (BI 201335 ZW) in plasma at steady state (CL/F,ss) following multiple oral administration
Time Frame: 10 minutes before drug administration and 1 hour (h),2h,3h,4h,5h,6h,8h,10h,11:50h, 23:50h on the last dose
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | BI 201335 NA Low TN | BI 201335 NA High TN | BI 201335 NA High TE
Number analyzed (Participants) | 5 | 6 | 6
mL/min | 28.2 (86.5) | 11.1 (68.0) | 8.01 (41.3)

ADVERSE EVENTS:
Time Frame: up to 72 weeks
Groups:
- Triple TN Placebo: Triple combination therapy for treatment naive patients- Patients receive a capsule containing matching placebo to BI 201335 NA (Placebo with IFN/RBV)
- Triple TN 120 mg: Triple combination therapy for treatment naive patients- Patients receive a capsule containing low dose of BI 201335 NA (120 mg q.d.) with IFN/RBV.
- Triple TN 240 mg: Triple combination therapy for treatment naive patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with IFN/RBV.
- Triple TE 240 mg: Triple combination therapy for treatment experienced patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with IFN/RBV.
- SOC TN Placebo: Standard of care for treatment naive patients- Patients receive a capsule containing matching placebo to BI 201335 NA (Placebo with IFN/RBV)
- SOC TN 120 mg: Standard of care for treatment naive patients- Patients receive a capsule containing low dose of BI 201335 NA (120 mg q.d.) with IFN/RBV.
- SOC TN 240 mg: Standard of care for treatment naive patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with IFN/RBV.
- SOC TE 240 mg: Standard of care for treatment experienced patients- Patients receive a capsule containing high dose of BI 201335 NA (240 mg q.d.) with IFN/RBV.
Arm/Group | Triple TN Placebo | Triple TN 120 mg | Triple TN 240 mg | Triple TE 240 mg | SOC TN Placebo | SOC TN 120 mg | SOC TN 240 mg | SOC TE 240 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 0/6 | 0/6 | 1/4 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 6/6 | 6/6 | 6/6 | 3/4 | 5/5 | 5/6 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triple TN Placebo (N=4) | Triple TN 120 mg (N=6) | Triple TN 240 mg (N=6) | Triple TE 240 mg (N=6) | SOC TN Placebo (N=4) | SOC TN 120 mg (N=5) | SOC TN 240 mg (N=6) | SOC TE 240 mg (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple TN Placebo (N=4) | Triple TN 120 mg (N=6) | Triple TN 240 mg (N=6) | Triple TE 240 mg (N=6) | SOC TN Placebo (N=4) | SOC TN 120 mg (N=5) | SOC TN 240 mg (N=6) | SOC TE 240 mg (N=6)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basedow's disease (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pingueculitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis atrophic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 1 | 2 | 1 | 0 | 3 | 2 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 4 | 1 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 1 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lymphocele (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.